CLINICAL TRIAL: NCT01390805
Title: Special Drug Use Investigation for VALTREX (Valaciclovir) (Suppression Prophylaxis)
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 112319
Record Dates: First submitted 2011-07-07; First posted 2011-07-11 (Estimated); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Genital Herpes
MeSH Terms: conditions — Herpes Genitalis | interventions — Valacyclovir

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Subjects with recurrent genital herpes
  Interventions: Drug: Valaciclovir Hydrochloride.

INTERVENTIONS:
Drug: Valaciclovir Hydrochloride.

SUMMARY:
The purpose of this study is to collect and assess information on proper use of valaciclovir regarding safety and efficacy of long-term use in suppressive therapy for subjects with recurrent genital herpes.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who started suppressive therapy for recurrent genital herpes for the first time

Exclusion Criteria:

* Subjects with a history of hypersensitivity to the ingredients of VALTREX or aciclovir

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Japanese subjects with recurrent genital herpes
Sampling Method: Probability Sample
Enrollment: 462 (Actual)
Dates: Start 2006-11; Primary Completion 2009-04 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
The number of adverse events in Japanese subjects with recurrent genital herpes treated with valaciclovir | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline